CLINICAL TRIAL: NCT01523977
Title: A Feasibility Trial of Everolimus (RAD001),an mTOR Inhibitor, Given in Combination With Multiagent Re-Induction Chemotherapy in Pediatric Patients With Relapsed Acute Lymphoblastic Leukemia (ALL)
Brief Title: Everolimus With Multiagent Re-Induction Chemotherapy in Pediatric Patients With ALL
Acronym: CRAD001NUS175T
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Lewis B. Silverman, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-237
Record Dates: First submitted 2012-01-30; First posted 2012-02-01 (Estimated); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: ALL; pediatric; relapse
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Recurrence | interventions — Everolimus; Prednisone; Vincristine; pegaspargase; Doxorubicin; Dexrazoxane

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Everolimus — Orally, daily days 1-32 per assigned dose level
  Other Names: RAD-001
Drug: Prednisone — 40 mg/m2/day orally 3 x daily days 4-32
Drug: Vincristine — 1.5 mg/m2 IV daily on days 4, 11, 18, and 25
Drug: PEG-Asparaginase — 2,500 U/m2 IV 1 x daily on days 5 and 18
  Other Names: Oncaspar
Drug: Doxorubicin — 30 mg/m2 IV on days 4 and 5
Drug: Dexrazoxane — 300 mg/m2 IV on days 4 and 5
  Other Names: Zinecard

SUMMARY:
Laboratory and other studies suggest that, the study drug, Everolimus (RAD001), may prevent tumor cell growth and also may increase the efficacy of other chemotherapy drugs. Everolimus is approved for use in the United States for certain types of cancer, such as kidney cancer. It has been extensively studied in people with various types of cancer as a single agent (a drug that is used alone to treat the cancer) or in combination with a number of other drugs. Studies in adults with cancer have also evaluated Everolimus in combination with other anti-tumor drugs. Information from lab studies and some other clinical trials suggests that Everolimus may kill leukemia cells on its own, and also make it more likely that steroids (such as prednisone) are able to kill leukemia cells.

In this research study, we are looking to learn more about how Everolimus works in combination with other drugs which are commonly used to treat relapsed acute lymphoblastic leukemia (prednisone, vincristine, PEG-asparaginase, and doxorubicin). The main goal of the study is to evaluate the side effects of this treatment combination in order to determine a safe dose of Everolimus which can be given with these other 4 drugs.

DETAILED DESCRIPTION:
Study Treatment: The study treatment lasts 32 days during which time you will be taking the study drug Everolimus daily for 32 days in addition to standard chemotherapy drugs. Below lists the study drug as well as the other drugs you will be receiving to treat your leukemia during this research study.

Chemotherapy drugs:

1. Everolimus (RAD001): By mouth Daily 1-32
2. Prednisone: By mouth or in the vein Three times daily on days 4-32
3. Vincristine: In the vein Daily on days 4, 11, 18, and 25
4. Doxorubicin: In the vein Once per day on days 4 and 5. A drug called dexrazoxane will be given with each dose of Doxorubicin to protect the heart from any damage that might be caused by Doxorubicin.
5. PEG-asparaginase: In the vein Once per day on days 5 and 18

If you have or have had an allergy to PEG-asparaginase, we will give another form of asparaginase (Erwinia asparaginase). Four doses of Erwinia asparaginase will be given in the muscle twice a week beginning on Day 5 and then another 4 doses will be given in the muscle twice a week beginning on Day 15 in place of the scheduled doses of PEG-asparaginase.

In addition to the medications listed above, you will also be receiving intrathecal (IT) chemotherapy that is given directly into your spinal fluid to treat the leukemia that may have spread to your brain and spinal fluid. The medicines we will be giving in your spinal fluid are listed below. The number of times we give chemotherapy into the spinal fluid will depend on whether or not we see leukemia cells in your spinal fluid on the sample we take on the first day of the study.

1. Cytarabine on Day 1 (also Day 4 if we see leukemia cells in your spinal fluid on the screening spinal tap)
2. Triple intrathecal therapy (cytarabine, methotrexate and hydrocortisone)on Days 18 and 32 (if we do not see leukemia cells in your spinal fluid on the screening spinal tap), or on Days 11, 18, 25 and 32 (if we see leukemia cells in your spinal fluid on the screening spinal tap)

A drug called leucovorin will be given by mouth or by vein after each dose of triple intrathecal therapy. Leucovorin is given to prevent mouth sores which might occur after you get methotrexate in the spinal fluid. Leucovorin will be given three times a day for 24 hours beginning one day after you receive a dose of triple intrathecal therapy.

Portions of this treatment are "routine" or "standard" ways of treating recurrent ALL. Receiving vincristine, prednisone, PEG asparaginase and doxorubicin along with chemotherapy in the spinal fluid is a standard treatment for relapsed leukemia. The research part of the treatment involves giving Everolimus at the same time as these drugs.

Clinical and Lab Exams: During the study, you will have a physical examinations and you will be asked questions about your general health and specific questions about any problems that you might be having and any medications you may be taking. You will also have blood work to check for any side effects to your organs from the study drug and other chemotherapy drugs. Bone marrow studies will be done at the end of the 32-day treatment period to assess how you responded to treatment. If you are in remission, a special minimal residual disease (MRD) test will also be performed from the marrow sample as part of the study.

ELIGIBILITY:
Inclusion Criteria:

* ALL in first bone marrow relapse occuring > 18 months from initial diagnosis
* Normal organ function
* Maximum prior cumulative doxorubicin dose of </= 360 mg/m2 or equivalent

Exclusion Criteria:

* Prior therapy for ALL except for intrathecal (IT) chemotherapy
* Pregnant or lactating
* Individuals whose relapsed ALL harbors a t(9;22)/BCR-ABL fusion
* Individuals whose lymphoblasts have surface immunoglobulin by flow cytometry and/or t(8;14), t(2;8), or t(8;22)
* Down syndrome
* Prior stem cell transplant
* History of asparaginase-associated pancreatitis
* Active lung disease
* Impairment of gastrointestinal function or gastrointestinal disease
* Severe and/or uncontrolled intercurrent illness
* Documented history of previous or current Hepatitis B or C infection
* History of a different malignancy (other than ALL) unless disease-free for at 5 years and deemed by the investigators to be at low risk for recurrence of that malignancy
* HIV positive on combination antiretroviral therapy

Ages: 18 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2011-11; Primary Completion 2017-01 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Safety and Feasibility | 2 years
  To determine the safety and feasibility of treatment with everolimus in combination with vincristine, prednisone, PEG-asparaginase and doxorubicin in patients with relapsed acute lymphoblastic leukemia (ALL)

SECONDARY OUTCOMES:
Clinical Activity | 2 years
  To investigate the clinical activity (complete remission rate and levels of end-reinduction MRD) of everolimus in combination with vincristine, prednisone, PEG-asparaginase and doxorubicin in patients with ALL.
Impact on biologic markers | 2 years
  To assess the impact of everolimus therapy when given in combination with vincristine, prednisone, PEG-asparaginase and doxorubicin on biologic markers of glucocorticoid resistance including levels of AKT, MCL1 and phosphorylated S6 ribosomal protein (PS6).
Determinants of Response | 2 years
  To explore possible determinants of response (as measured by peripheral blast clearance, MRD levels and CR status) to everolimus in combination with multi-agent therapy including measurements of anti-apoptotic proteins (BCL2, BCLxL and MCL1), genome-wide gene expression profliling, BH3 profiling and OncoMap profiling.

CONTACTS AND LOCATIONS:
Overall Officials: Lewis Silverman, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (8):
- United States (8):
  - UCSF, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Boston Children's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Columbia University Medical Center, New York, New York
  - Seattle Children's Hospital, Seattle, Washington